CLINICAL TRIAL: NCT03771963
Title: An Open-Label, Phase 3 Trial to Investigate the Immunogenicity and Safety of Tetravalent Dengue Vaccine Candidate (TDV) at the End of Shelf Life in Healthy Adults in Non-Endemic Country(Ies) for Dengue
Brief Title: Immunogenicity and Safety of Tetravalent Dengue Vaccine (TDV) at the End of Shelf Life in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DEN-307; U1111-1222-2812 (Registry Identifier: WHO)
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Dengue Fever
Keywords: Live Attenuated Tetravalent Dengue Vaccine
MeSH Terms: conditions — Dengue | interventions — Dengue Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tetravalent Dengue Vaccine (TDV) (Experimental): TDV 0.5 mL, injection, subcutaneously (SC), once on Day 1 (first dose) and Day 90 (second dose).
  Interventions: Biological: Tetravalent Dengue Vaccine (TDV)

INTERVENTIONS:
Biological: Tetravalent Dengue Vaccine (TDV) — TDV SC injection.

SUMMARY:
The purpose of this study is to evaluate the safety and immune response of a naturally aged lot of tetravalent dengue vaccine (TDV) in healthy participants, aged 18 to 60 years, in non-endemic country(ies) for dengue.

DETAILED DESCRIPTION:
The vaccine being tested in this study is tetravalent dengue vaccine (TDV). The primary objective of this study is to evaluate the immune response and safety of a naturally aged (>12 months stored at 2°C to 8°C) lot of TDV in a healthy adult population in country(ies) non-endemic for dengue. The assessment of a naturally aged lot of TDV in this clinical trial will provide an important contribution to data on TDV stability throughout the shelf life of the product.

The study will enroll approximately 200 participants. Participants will be enrolled to the one treatment group:

Tetravalent Dengue Vaccine (TDV)

All participants will receive subcutaneous (SC) injection on Day 1 (Month 0) and Day 90 (Month 3).

This multi-center trial will be conducted in the United States. The overall time to participate in this study is 9 months. Participants will make multiple visits to the clinic including a final visit at Day 270 (Month 9).

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs), and the clinical judgment of the investigator.
2. Participants who sign and date a written informed consent form and any required privacy authorization prior to the initiation of any trial procedures, after the nature of the trial has been explained according to local regulatory requirements.

Exclusion Criteria:

1. Participants with a clinically significant active infection (as assessed by the investigator) or body temperature ≥38°C (≥100.4°F) within 3 days of the intended date of vaccine administration
2. Known or suspected impairment/alteration of immune function, including:

   1. Chronic use of oral steroids (equivalent to 20 mg/day prednisone ≥12 weeks and/or ≥2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (Month 0) (use of inhaled, intranasal, or topical corticosteroids is allowed).
   2. Receipt of parenteral steroids (equivalent to 20 mg/day prednisone ≥12 weeks and/or ≥2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (Month 0).
   3. Administration of immunoglobulins and/or any blood products within the 3 months prior to Day 1 (Month 0) or planned administration during the trial.
   4. Receipt of immunostimulants within 60 days prior to Day 1 (Month 0).
   5. Immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within 6 months prior to Day 1 (Month 0).
   6. Known Human Immunodeficiency Virus (HIV) infection or HIV-related disease.
   7. Hepatitis C virus infection.
   8. Genetic immunodeficiency.
3. With Body Mass Index (BMI) greater than or equal to 35 kg/m^2(=weight in kg/height in meters^2).
4. Participants who have known hypersensitivity or allergy to any of the vaccine components.
5. Previous and planned vaccination (during the trial conduct), against any flavivirus including dengue, Yellow Fever (YF), Japanese Encephalitis (JE) viruses or tick-borne encephalitis.
6. Previous participation in any clinical trial of a dengue or other flavivirus (e.g., West Nile [WN] virus) candidate vaccine, except for participants who received placebo in those trials.
7. With a current or previous infection with a flavivirus such as dengue, Zika, YF, JE, WN fever, tick-borne encephalitis or Murray Valley encephalitis and participants with a history of prolonged (≥1 year) habitation in a dengue endemic area.
8. Participants with any history of progressive or severe neurologic disorder, seizure disorder or neuro-inflammatory disease (e.g., Guillain-Barré syndrome).
9. Participants with history of substance or alcohol abuse within the past 2 years.
10. Participants who have any serious chronic or progressive disease according to judgment of the Investigator (e.g., neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- United States (2):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Hutchinson Clinic, Hutchinson, Kansas

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Rauscher M, Youard Z, Faccin A, Patel SS, Pang H, Zent O. Pregnancy outcomes following unintentional exposure to TAK-003, a live-attenuated tetravalent dengue vaccine. Expert Rev Vaccines. 2025 Dec;24(1):221-229. doi: 10.1080/14760584.2025.2480297. Epub 2025 Mar 27. PMID 40099800
- [Derived] Patel SS, Winkle P, Faccin A, Nordio F, LeFevre I, Tsoukas CG. An open-label, Phase 3 trial of TAK-003, a live attenuated dengue tetravalent vaccine, in healthy US adults: immunogenicity and safety when administered during the second half of a 24-month shelf-life. Hum Vaccin Immunother. 2023 Aug;19(2):2254964. doi: 10.1080/21645515.2023.2254964. Epub 2023 Oct 17. PMID 37846724

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 28 March 2019 to 13 March 2020.
Pre-assignment Details: Healthy participants were enrolled in this study to receive Tetravalent Dengue Vaccine (TDV) on Days 1 and 90.
Period: Overall Study
Arm/Group | Tetravalent Dengue Vaccine (TDV)
Started | 200
Completed | 168
Not Completed | 32
Not completed — Lost to Follow-up | 22
Not completed — Withdrawal of Consent | 10

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who received at least 1 dose of TDV trial vaccine.
Arm/Group | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.27 (12.035)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 64
  Not Hispanic or Latino | 136
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 41
  White | 148
  More than one race | 3
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 200
Height [Mean (Standard Deviation); unit: cm] | 170.72 (9.330)
Weight [Mean (Standard Deviation); unit: kg] | 80.23 (15.220)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI= weight (kg)/[height (m)^2]
  kg/m^2 | 27.45 (4.248)

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMT) of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at Day 120
Description: GMTs of neutralizing antibodies for each of the 4 dengue serotypes were measured by microneutralization test 50% [MNT50]. The 4 dengue virus serotypes were DENV-1, DENV-2, DENV-3, and DENV-4.
Time Frame: One month post second dose (Day 120)
Population: Per-protocol Set (PPS) excludes all participants seropositive for dengue virus at Baseline and includes all participants in the Full Analysis Set (FAS- who received at least 1 dose of trial vaccine with valid pre-dose and post-dose measurement for immunogenicity assessment) who have no major protocol violations, with data available for analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 132
titer
  DENV-1 | 557.4 [417.0 to 744.9]
  DENV-2 | 2047.4 [1739.7 to 2409.5]
  DENV-3 | 131.8 [105.0 to 165.4]
  DENV-4 | 119.6 [97.7 to 146.5]

2. Secondary Outcome: Seropositivity Rates for Each of the 4 Dengue Serotypes at Days 120 and 270
Description: Seropositivity rate was defined as the percentage of participants being seropositive, derived from titers of dengue-neutralizing antibodies. Seropositivity was defined as a reciprocal neutralizing titer ≥10 (for each serotype). Seropositivity rates were assessed for the four dengue serotypes: DENV-1, DENV-2, DENV-3, and DENV-4.
Time Frame: One month and six months post second dose (Days 120 and 270)
Population: The PPS excludes all participants seropositive for dengue virus at Baseline and includes all participants in the FAS who have no major protocol violations. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 139
percentage of participants
  Day 120: DENV-1: number analyzed (Participants) | 132
  Day 120: DENV-1 | 99.2 [95.9 to 100.0]
  Day 120: DENV-2: number analyzed (Participants) | 132
  Day 120: DENV-2 | 100.0 [97.2 to 100.0]
  Day 120: DENV-3: number analyzed (Participants) | 132
  Day 120: DENV-3 | 97.7 [93.5 to 99.5]
  Day 120: DENV-4: number analyzed (Participants) | 132
  Day 120: DENV-4 | 99.2 [95.9 to 100.0]
  Day 270: DENV-1: number analyzed (Participants) | 133
  Day 270: DENV-1 | 97.0 [92.5 to 99.2]
  Day 270: DENV-2: number analyzed (Participants) | 133
  Day 270: DENV-2 | 98.5 [94.7 to 99.8]
  Day 270: DENV-3: number analyzed (Participants) | 133
  Day 270: DENV-3 | 85.7 [78.6 to 91.2]
  Day 270: DENV-4: number analyzed (Participants) | 133
  Day 270: DENV-4 | 86.5 [79.5 to 91.8]

3. Secondary Outcome: Seropositivity Rates for Multiple (2, 3, or 4) Dengue Serotypes at Days 120 and 270
Description: Seropositivity rate was defined as the percentage of participants being seropositive, derived from titers of dengue-neutralizing antibodies. Seropositivity was defined as a reciprocal neutralizing titer ≥10. The dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Seropositivity for multiple dengue serotypes was summarized in the following categories: tetravalent and at least trivalent.
Time Frame: One month and six months post second dose (Days 120 and 270)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 139
percentage of participants
  Day 120: At Least Trivalent: number analyzed (Participants) | 132
  Day 120: At Least Trivalent | 99.2 [95.9 to 100.0]
  Day 120: Tetravalent: number analyzed (Participants) | 132
  Day 120: Tetravalent | 97.0 [92.4 to 99.2]
  Day 270: At Least Trivalent: number analyzed (Participants) | 133
  Day 270: At Least Trivalent | 91.0 [84.8 to 95.3]
  Day 270: Tetravalent: number analyzed (Participants) | 133
  Day 270: Tetravalent | 78.9 [71.0 to 85.5]

4. Secondary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at Day 270
Description: GMTs of neutralizing antibodies were assessed for the four dengue serotypes: DENV-1, DENV-2, DENV-3, and DENV-4, by MNT50.
Time Frame: Six months post second dose (Day 270)
Population: PPS excludes all participants seropositive for dengue virus at Baseline and includes all participants in the FAS who have no major protocol violations, with data available for analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 133
titer
  DENV-1 | 311.6 [222.8 to 435.9]
  DENV-2 | 1170.6 [953.9 to 1436.5]
  DENV-3 | 63.0 [48.4 to 82.0]
  DENV-4 | 57.6 [44.2 to 75.0]

5. Secondary Outcome: Percentage of Participants With Solicited Local (Injection Site) Reactions Following Each Vaccination by Severity
Description: Solicited local adverse events (AEs) [at injection site] were collected by participants using diary cards within 7 days after each vaccination and included injection site pain [Grade 0 (no pain), 1 (mild: no interference with daily activity), 2 (moderate: interference with daily activity with or without treatment) and 3 (severe: prevents daily activity with or without treatment)], injection site erythema [Grade 0 (<25 mm), 1 (25 - ≤ 50 mm), 2 (>50 - ≤ 100 mm), 3 (> 100 mm)] and injection site swelling [Grade 0 (<25 mm), 1 (25 - ≤ 50 mm), 2 (>50 - ≤ 100 mm), 3 (> 100 mm)]. The percentages were rounded off to the first decimal place. Only categories with at least 1 participant are reported.
Time Frame: Up to 7 days (Day of vaccination + 6 subsequent days) after each of the vaccination
Population: Safety Set included all participants who received at least 1 dose of TDV trial vaccine. Number analyzed is the number of participants with data available for the specific category.
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 200
percentage of participants
  After First Vaccination, Any Solicited Local AEs: number analyzed (Participants) | 192
  After First Vaccination, Any Solicited Local AEs | 35.9
  After First Vaccination, Pain: Any Severity: number analyzed (Participants) | 192
  After First Vaccination, Pain: Any Severity | 29.7
  After First Vaccination, Pain: Mild: number analyzed (Participants) | 192
  After First Vaccination, Pain: Mild | 25.5
  After First Vaccination, Pain: Moderate: number analyzed (Participants) | 192
  After First Vaccination, Pain: Moderate | 3.6
  After First Vaccination, Pain: Severe: number analyzed (Participants) | 192
  After First Vaccination, Pain: Severe | 0.5
  After First Vaccination, Erythema: Any Severity: number analyzed (Participants) | 192
  After First Vaccination, Erythema: Any Severity | 13.0
  After First Vaccination, Erythema: Mild: number analyzed (Participants) | 192
  After First Vaccination, Erythema: Mild | 12.0
  After First Vaccination, Erythema: Moderate: number analyzed (Participants) | 192
  After First Vaccination, Erythema: Moderate | 1.0
  After First Vaccination, Swelling: Any Severity: number analyzed (Participants) | 192
  After First Vaccination, Swelling: Any Severity | 4.2
  After First Vaccination, Swelling: Mild: number analyzed (Participants) | 192
  After First Vaccination, Swelling: Mild | 4.2
  After Second Vaccination, Any Solicited Local AEs: number analyzed (Participants) | 167
  After Second Vaccination, Any Solicited Local AEs | 32.3
  After Second Vaccination, Pain: Any Severity: number analyzed (Participants) | 167
  After Second Vaccination, Pain: Any Severity | 31.1
  After Second Vaccination, Pain: Mild: number analyzed (Participants) | 167
  After Second Vaccination, Pain: Mild | 27.5
  After Second Vaccination, Pain: Moderate: number analyzed (Participants) | 167
  After Second Vaccination, Pain: Moderate | 2.4
  After Second Vaccination, Pain: Severe: number analyzed (Participants) | 167
  After Second Vaccination, Pain: Severe | 1.2
  After Second Vaccination, Erythema: Any Severity: number analyzed (Participants) | 167
  After Second Vaccination, Erythema: Any Severity | 6.0
  After Second Vaccination, Erythema: Mild: number analyzed (Participants) | 167
  After Second Vaccination, Erythema: Mild | 6.0
  After Second Vaccination, Swelling: Any Severity: number analyzed (Participants) | 167
  After Second Vaccination, Swelling: Any Severity | 2.4
  After Second Vaccination, Swelling: Mild: number analyzed (Participants) | 167
  After Second Vaccination, Swelling: Mild | 2.4

6. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events Following Each Vaccination by Severity
Description: Solicited systemic AEs were collected by participants using diary cards within 14 days after each vaccination and included fever, headache, asthenia, malaise and myalgia. Severity grades were: Grade 0: none, Grade 1: mild (no interference with daily activity), Grade 2: moderate (interference with daily activity with or without treatment), Grade 3: severe (prevents normal daily activity with or without treatment). Fever is defined as body temperature greater than or equal to 38°C (100.4°F). Fever was excluded from the overall count as no severity grading was applied for it. The percentages were rounded off to the first decimal place. Only categories with at least 1 participant are reported.
Time Frame: Up to 14 days (Day of vaccination + 13 subsequent days) after each vaccination
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 200
percentage of participants
  After First Vaccination, Any Solicited Systemic Local AEs: number analyzed (Participants) | 192
  After First Vaccination, Any Solicited Systemic Local AEs | 42.2
  After First Vaccination, Headache: Any Severity: number analyzed (Participants) | 192
  After First Vaccination, Headache: Any Severity | 30.2
  After First Vaccination, Headache: Mild: number analyzed (Participants) | 192
  After First Vaccination, Headache: Mild | 22.9
  After First Vaccination, Headache: Moderate: number analyzed (Participants) | 192
  After First Vaccination, Headache: Moderate | 5.7
  After First Vaccination, Headache: Severe: number analyzed (Participants) | 192
  After First Vaccination, Headache: Severe | 1.6
  After First Vaccination, Myalgia: Any Severity: number analyzed (Participants) | 192
  After First Vaccination, Myalgia: Any Severity | 25.5
  After First Vaccination, Myalgia: Mild: number analyzed (Participants) | 192
  After First Vaccination, Myalgia: Mild | 20.8
  After First Vaccination, Myalgia: Moderate: number analyzed (Participants) | 192
  After First Vaccination, Myalgia: Moderate | 3.1
  After First Vaccination, Myalgia: Severe: number analyzed (Participants) | 192
  After First Vaccination, Myalgia: Severe | 1.6
  After First Vaccination, Asthenia: Any Severity: number analyzed (Participants) | 192
  After First Vaccination, Asthenia: Any Severity | 16.7
  After First Vaccination, Asthenia: Mild: number analyzed (Participants) | 192
  After First Vaccination, Asthenia: Mild | 10.4
  After First Vaccination, Asthenia: Moderate: number analyzed (Participants) | 192
  After First Vaccination, Asthenia: Moderate | 5.2
  After First Vaccination, Asthenia: Severe: number analyzed (Participants) | 192
  After First Vaccination, Asthenia: Severe | 1.0
  After First Vaccination, Malaise: Any Severity: number analyzed (Participants) | 192
  After First Vaccination, Malaise: Any Severity | 19.8
  After First Vaccination, Malaise: Mild: number analyzed (Participants) | 192
  After First Vaccination, Malaise: Mild | 13.0
  After First Vaccination, Malaise: Moderate: number analyzed (Participants) | 192
  After First Vaccination, Malaise: Moderate | 4.7
  After First Vaccination, Malaise: Severe: number analyzed (Participants) | 192
  After First Vaccination, Malaise: Severe | 2.1
  After First Vaccination, Fever: Any: number analyzed (Participants) | 189
  After First Vaccination, Fever: Any | 2.6
  After First Vaccination, Fever: 38.0-<38.5: number analyzed (Participants) | 189
  After First Vaccination, Fever: 38.0-<38.5 | 2.1
  After First Vaccination, Fever: 38.5-<39.0: number analyzed (Participants) | 189
  After First Vaccination, Fever: 38.5-<39.0 | 0.5
  After Second Vaccination, Any Solicited Systemic Local AEs: number analyzed (Participants) | 167
  After Second Vaccination, Any Solicited Systemic Local AEs | 34.1
  After Second Vaccination, Headache: Any Severity: number analyzed (Participants) | 167
  After Second Vaccination, Headache: Any Severity | 22.8
  After Second Vaccination, Headache: Mild: number analyzed (Participants) | 167
  After Second Vaccination, Headache: Mild | 16.2
  After Second Vaccination, Headache: Moderate: number analyzed (Participants) | 167
  After Second Vaccination, Headache: Moderate | 5.4
  After Second Vaccination, Headache: Severe: number analyzed (Participants) | 167
  After Second Vaccination, Headache: Severe | 1.2
  After Second Vaccination, Myalgia: Any Severity: number analyzed (Participants) | 167
  After Second Vaccination, Myalgia: Any Severity | 22.2
  After Second Vaccination, Myalgia: Mild: number analyzed (Participants) | 167
  After Second Vaccination, Myalgia: Mild | 20.4
  After Second Vaccination, Myalgia: Moderate: number analyzed (Participants) | 167
  After Second Vaccination, Myalgia: Moderate | 1.2
  After Second Vaccination, Myalgia: Severe: number analyzed (Participants) | 167
  After Second Vaccination, Myalgia: Severe | 0.6
  After Second Vaccination, Asthenia: Any Severity: number analyzed (Participants) | 167
  After Second Vaccination, Asthenia: Any Severity | 12.0
  After Second Vaccination, Asthenia: Mild: number analyzed (Participants) | 167
  After Second Vaccination, Asthenia: Mild | 7.8
  After Second Vaccination, Asthenia: Moderate: number analyzed (Participants) | 167
  After Second Vaccination, Asthenia: Moderate | 3.0
  After Second Vaccination, Asthenia: Severe: number analyzed (Participants) | 167
  After Second Vaccination, Asthenia: Severe | 1.2
  After Second Vaccination, Malaise: Any Severity: number analyzed (Participants) | 167
  After Second Vaccination, Malaise: Any Severity | 13.2
  After Second Vaccination, Malaise: Mild: number analyzed (Participants) | 167
  After Second Vaccination, Malaise: Mild | 9.0
  After Second Vaccination, Malaise: Moderate: number analyzed (Participants) | 167
  After Second Vaccination, Malaise: Moderate | 3.0
  After Second Vaccination, Malaise: Severe: number analyzed (Participants) | 167
  After Second Vaccination, Malaise: Severe | 1.2
  After Second Vaccination, Fever: Any: number analyzed (Participants) | 166
  After Second Vaccination, Fever: Any | 1.2
  After Second Vaccination, Fever: 38.0-<38.5: number analyzed (Participants) | 166
  After Second Vaccination, Fever: 38.0-<38.5 | 0.6
  After Second Vaccination, Fever: 38.5-<39.0: number analyzed (Participants) | 166
  After Second Vaccination, Fever: 38.5-<39.0 | 0.6

7. Secondary Outcome: Percentage of Participants With Any Unsolicited Adverse Events Following Each Vaccination
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a study vaccine; it does not necessarily have to have a causal relationship with study vaccine administration.
Time Frame: Up to 28 days after each vaccination (Day of vaccination + 27 subsequent days)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 200
percentage of participants
  After First Vaccination | 11.5
  After Second Vaccination: number analyzed (Participants) | 176
  After Second Vaccination | 10.8

8. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, leads to a congenital anomaly / birth defect in the offspring of a participant, or is an important medical event which may require intervention to prevent the items listed above or may expose the participant to danger, even though the event is not immediately life threatening or fatal or does not result in hospitalization.
Time Frame: From first vaccination (Day 1) through end of study (Day 270)
Population: Safety Set included all participants who received at least 1 dose of TDV trial vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 200
percentage of participants | 2.5

9. Secondary Outcome: Percentage of Participants With Medically Attended Adverse Events (MAAEs)
Description: MAAEs are defined as AEs leading to an unscheduled visit to or by a healthcare professional, including visits to an emergency department, but not fulfilling seriousness criteria.
Time Frame: From first vaccination (Day 1) through end of study (Day 270)
Population: Safety Set included all participants who received at least 1 dose of TDV trial vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Dengue Vaccine (TDV)
Number analyzed (Participants) | 200
percentage of participants | 26.0

ADVERSE EVENTS:
Time Frame: All-cause mortality and Serious adverse events: From first vaccination (Day 1) through end of study (Day 270). Other (Non-serious) adverse events: Up to 28 days after each vaccination (Day of vaccination + 27 subsequent days).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Tetravalent Dengue Vaccine (TDV)
All-Cause Mortality (participants affected / at risk) | 0/200
Serious Adverse Events (participants affected / at risk) | 5/200
Other Adverse Events (participants affected / at risk) | 0/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tetravalent Dengue Vaccine (TDV) (N=200)
Bradycardia (Cardiac disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Sepsis (Infections and infestations) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/63/NCT03771963/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT03771963/SAP_001.pdf